CLINICAL TRIAL: NCT06446466
Title: Influence of Pulsed Electromagnetic Fields (PEMFs) Stimulation on Physical Exercise in Sedentary People
Brief Title: PEMF Stimulation on Physical Exercise in Sedentary People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Milena Raffi, Associate professor, University of Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PEMF on sedentary
Record Dates: First submitted 2024-05-03; First posted 2024-06-06 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: PEMF Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants group (Experimental): Two interventions will be performed on the same group of subjects. Participants will be healthy volunteers with sedentary habits.
  The experiments will be performed on the cycle-ergometer (H-300-R Lode, Exere Air Machine, Italy). The surface EMG activity will be recorded from the right Vastus Medialis and right Biceps Femoris caput longum at a sampling rate of 1000 Hz by a Free-EMG 1000 (BTS Bioengineering, Inc.). To stimulate the entire right thigh, 2 circular 20 cm PEMF loop-antenna devices (Torino II, Rio Grande Neurosciences, USA) will be placed at the beginning and at the end of the right leg. The PEMF waveform consists of a pulse-burst modulated 27.12 Mega-Hertz (MHz) sinusoidal carrier, with 2ms burst width repeated at 2 Hertz, with peak magnetic field at the center of the loop 5±1 microTesla.
  Interventions: Device: PEMF ON-OFF; Device: PEMF OFF-ON

INTERVENTIONS:
Device: PEMF ON-OFF — In the experimental condition PEMF ON-OFF, the participants will start the exercise session with PEMF in ON modality. The PEMF device will be kept ON for 17 minutes. Then, it will be turned OFF while the participant will keep going cycling until the end of the trial.
  This condition is used to investigate the effect on PEMF at the onset of the exercise. Data acquired in the first 17 minutes (PEMF ON) will be compared with those recorded in the last 17 minutes (PEMF OFF) of the exercise session.
Device: PEMF OFF-ON — In the experimental condition PEMF OFF-ON, the participants will start the exercise session with PEMF in OFF modality. The PEMF device will be kept OFF for 17 minutes. Then, it will be turned ON and the participant will keep going cycling until the end of the trial.
  This condition is used to investigate the effect of PEMF during the exercise, when the muscle will have worked for 17 minutes. Data acquired in the first 17 minutes (PEMF OFF) will be compared with those recorded in the last 17 minutes (PEMF ON) of the exercise session.

SUMMARY:
The pulsed electromagnetic fields (PEMF) are a non-invasive therapy used for clinical treatments. Recent publications in exercise physiology showed that PEMF enhanced the velocity and the quantity of available muscle O2, and the rate of muscle oxygen extraction and utilization, in semi-professional cyclists during a heavy constant-load exercise. This study investigates the effect of stimulation on muscular activation in sedentary young people who perform a constant-load exercise at moderate intensity. The protocols foresees the enrollment of nine male sedentary young people. The response of the muscle activity will be recorded by surface electromyography (EMG) and assessed by measuring the root mean square normalized to the peak of the maximum voluntary contraction. Data will be collected in the vastus Medialis (RVM) and Biceps Femoris (RBF) of the right leg, at the baseline (standstill sitting), on warm-up (unloaded cy-cling) and during 30 minutes of constant-load exercise in two experimental conditions (PEMF ON vs PEMF OFF).

DETAILED DESCRIPTION:
The study design is single-blind with randomized controlled condition. Nine male sedentary young people will participate at this study. G∗power software version 3.1.9.2 (Kiel, Germany) predicted that a total sample size of 8 would give sufficient power (0.80) to detect a significant difference at alpha level of 0.05. One additional participant will be included to ensure the availability of data in case of missing or corrupted data. All participants will be volunteers, healthy, non-smokers, without muscular injury or physical deficit at the time of the experiment. Exclusion criteria are the use of supplements or medications. All participants will receive both a written and verbal explanation of the experimental procedure. The informed consent will be obtained before the beginning of recordings.

The experiments will be performed on the cycle-ergometer (H-300-R Lode, Exere Air Machine, Italy) under a standardized procedure in a quiet room with a temperature of 22°C. Recordings will be performed at the same time of the day (9:00-12:00 AM) to avoid circadian influence. Subjects will be instructed to avoid caffeine, alcohol and heavy physical activity in the 12h preceding the experiment. The surface EMG activity will be recorded from the right Vastus Medialis and right Biceps Femoris caput longum at a sampling rate of 1000 Hz by a Free-EMG 1000 (BTS Bioengineering, Inc.). Free-EMG is a device with wireless miniaturized probes for the dynamic analysis of muscle activity. For signal acquisition, the probes (41,5×24,8x14mm) are directly attached to the electrodes and signals are detected and captured. Each probe is equipped with internal memory to ensure uninterrupted recording in case of temporary connection loss. To stimulate the entire right thigh, 2 circular 20 cm PEMF loop-antenna devices (Torino II, Rio Grande Neurosciences, USA) will be placed at the beginning and at the end of the right leg. The PEMF waveform consists of a pulse-burst modulated 27.12 Mega-Hertz (MHz) sinusoidal carrier, with 2ms burst width repeated at 2 Hertz, with peak magnetic field at the center of the loop 5±1 microTesla.

Participants will come to the laboratory 5 times, with an interval of 3 days between each time. In each of these visits few recordings will be performed.

The first day foresees the recording of the maximum voluntary contraction (MVC) and an incremental test until exhaustion to find the individual maximum oxygen consumption (VO2max). Regarding MVC recording, each participant will perform, for five seconds, an isometric contraction against a maximum load using isotonic machines (Exere Air Machine, Italy). The participants will repeat the same procedure 3 times, separated by 2 minutes of rest. The MVC peak value of each investigated muscle will be used to normalize electromyographic data (procedure already used in previous studies). Regarding VO2max recording, each subject will perform an incremental test on a cycle-ergometer (H-300-R Lode) to find the maximum oxygen consumption (VO2max), in order to individualize the correct workload to be used for the exercise sessions. Gases will be analyzed using a Quark b2 breath-by-breath metabolic system (Cosmed, Italy). The system will be calibrated immediately before each test in accordance with the manufacturer's guidelines: volume calibration will be performed at different flow rates with a 3- L calibration syringe and calibration of gas analyzers will be performed with a tank of reference gas mixture (16.00% O2, 5.00% CO2) and ambient air (20.93% O2 and 0.03% CO2).

From day two to four, participants will come to the laboratory for the exercise sessions. The experimental conditions will be PEMF ON and PEMF OFF, in which the PEMF will be turned on and off respectively. When the trial will start with the PEMF in ON modality, the device will be turned off after 17 minutes and the participant will keep going cycling until the end of the trial. Otherwise, when the trial will start with the PEMF in OFF modality, the device will be turned on after 17 minutes and the participant will keep going cycling until the end of the trial. Each condition will be repeated twice in different days for a total of four recordings per subject. The two PEMF loops will be positioned on the right leg in both experimental conditions in order to avoid stimulation being perceived by the subjects at the skin level.

Data will be recorded in three epochs: 1) baseline, 2) warm-up, 3) constant-load exercise. To record the baseline values, the participants will sit for 1-minute with the right leg extended. The warm-up involves an unloaded cycling for 1-minute. Then, an instantaneous increase of the workload, which will be attained in ~3s, will be the onset for the constant-load exercise (physical effort). Participants will be instructed to keep cycling at a cadence of 70 revolutions per minute for the entire duration of the trial. Each trial will be ended after 30 minutes of exercise.

ELIGIBILITY:
Inclusion Criteria:

- healthy sedentary volunteers

Exclusion Criteria:

* smokers
* muscular injury or physical deficit at the time of the experiment
* use of supplements or medications

Ages: 23 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-11-12 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-02-03 (Actual)

PRIMARY OUTCOMES:
PEMF effect on amplitude of muscle contraction | Two weeks recordings
  The aim is to verify if PEMF stimulation can enhance muscle activity during cycling. Electromyographic recordings on both vastus Medialis (RVM) and Biceps Femoris (RBF) of the right leg will be performed. To verify the effect, the amplitude (in mV) of the muscle response will be analyzed.
PEMF effect on duration of muscle contraction | Two weeks recordings
  The aim is to verify if PEMF stimulation can enhance muscle activity during cycling. Electromyographic recordings on both vastus Medialis (RVM) and Biceps Femoris (RBF) of the right leg will be performed. To verify the effect, the duration (in msec) of the muscle response will by analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Milena Raffi, PhD, Principal Investigator — University of Bologna
Locations (1):
- Record Sport - Via del Pilastro 8, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trofe A, Piras A, Muehsam D, Meoni A, Campa F, Toselli S, Raffi M. Effect of Pulsed Electromagnetic Fields (PEMFs) on Muscular Activation during Cycling: A Single-Blind Controlled Pilot Study. Healthcare (Basel). 2023 Mar 22;11(6):922. doi: 10.3390/healthcare11060922. PMID 36981580
- [Background] Raffi M, Piras A, Persiani M, Perazzolo M, Squatrito S. Angle of gaze and optic flow direction modulate body sway. J Electromyogr Kinesiol. 2017 Aug;35:61-68. doi: 10.1016/j.jelekin.2017.05.008. Epub 2017 May 31. PMID 28601564